CLINICAL TRIAL: NCT01714375
Title: Daily Exposure Monitoring of Noise Study
Brief Title: Daily Exposure Monitoring to Prevent Hearing Loss
Acronym: DEMON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0509000588; 1R01OH008641-01 (NIH)
Record Dates: First submitted 2012-10-22; First posted 2012-10-25 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- QuietDose device VOLUNTARY (Active Comparator): This group of employees will voluntarily use the "QuietDose" units in place of their regular hearing protection, which may be either ear plugs or ear muffs.
  Interventions: Device: QuietDose Device
- No QuietDose device (No Intervention): This group of employees will not use the "QuietDose" units and maintain use of their regular hearing protection which may be either ear plugs or ear muffs.
- QuietDose Device REQUIRED (Active Comparator): This group of employees will be required to use the "QuietDose" units in place of their regular hearing protection, which may be either ear plugs or ear muffs.
  Interventions: Device: QuietDose Device

INTERVENTIONS:
Device: QuietDose Device — The intervention will test the effectiveness of a noise exposure dosimeter, the QuietDose - that measures a worker's daily noise "dose", as well as peak noise exposure, inside of the worker's hearing protectors. Workers and the study coordinator receive daily feedback about noise exposures (if the device was used outside of the study it would be safety personnel that received the feedback outside of the workers themselves). Such feedback will allow steps to be taken to minimize such exposures, such as behavioral adjustments and improved awarenessThe goal of this study is to determine whether daily assessment and feedback of workers' noise exposures leads to more effective use of hearing protection and prevention of noise-induced hearing loss.
  Arms: QuietDose Device REQUIRED; QuietDose device VOLUNTARY

SUMMARY:
The goal of this study is to determine whether daily assessment and feedback of workers' noise exposures leads to more effective use of hearing protection and prevention of noise-induced hearing loss.

DETAILED DESCRIPTION:
Despite the existence of an OSHA standard for hearing conservation, noise-induced hearing loss continues to be one of the most prevalent occupational conditions. Furthermore, hearing loss rates appear to vary significantly between industrial locations with similar measured noise exposure levels. The factors that determine an effective hearing conservation program remain poorly understood. The effective use of hearing protection, believed to be a critical component of such programs, is felt to be highly variable in real world situations. Provocative new data by our research group indicate that much of the preventable hearing loss in a large industrial workforce is occurring not among the workers in the highest ambient noise areas, but instead among employees working in areas where measured ambient median noise exposures are close to or even slightly below the current OSHA action level (85dBA for an 8 hour time weighted average). One possible reason could be that the use of hearing protection is currently less effective in such areas of lower or intermittent noise compared to high noise areas. Since in many worksites, the majority of workers are exposed to moderate noise levels, there is an urgent need to better understand how to prevent hearing loss in these settings. There are also currently no national guidelines for ensuring correct fit and function of hearing protection, and there is an urgent need to find ways to promote the correct use of hearing protective devices. This study will assess the impact of hearing protector fit testing and daily noise exposure monitoring, with major implications for hearing conservation practice, and the wider prevention of noise-induced hearing loss. It will also explore the role of hearing protective devices in areas of median noise exposure less than 85dBA.

This proposed study is a worksite intervention trial of a new technology to reduce occupational noise-induced hearing loss. The intervention will test the effectiveness of a noise exposure dosimeter, the QuietDose - essentially a small microphone connected to a noise logging device about the size of a beeper- that measures a worker's daily noise "dose", as well as peak noise exposure, inside of the worker's hearing protectors. Workers and the study coordinator receive daily feedback about noise exposures (if the device was used outside of the study it would be safety personnel that received the feedback outside of the workers themselves). Such feedback will allow steps to be taken to minimize such exposures, such as behavioral adjustments and improved awarenessThe goal of this study is to determine whether daily assessment and feedback of workers' noise exposures leads to more effective use of hearing protection and prevention of noise-induced hearing loss. The proposed study will take advantage of the unique working relationship between a research institution (the Yale Occupational and Environmental Medicine Program) and a major industrial corporation (Alcoa, Inc.) to conduct this intervention trial at several of the company's facilities.

ELIGIBILITY:
Inclusion Criteria:

The only criterion for inclusion is that the employee is currently working in an area where there is sufficient noise exposure that the company's policy requires the use of hearing protection.

Exclusion Criteria:

There are no exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2007-07-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Hearing Loss | 1 year
  Hearing loss will be measured in dB/year for the noise-sensitive audiometric frequency averages of 2, 3, and 4000 Hz and 3, 4, and 6000 Hz averaged across ears .

CONTACTS AND LOCATIONS:
Overall Officials: Peter M Rabinowitz, MD MPH, Principal Investigator — Yale Occupational and Environmental Medicine Program: Yale University School of Medicine
Locations (1):
- Yale Occupational and Environmental Medicine Program, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Rabinowitz P, Galusha D, Cantley LF, Dixon-Ernst C, Neitzel R. Feasibility of a daily noise monitoring intervention for prevention of noise-induced hearing loss. Occup Environ Med. 2021 Nov;78(11):835-840. doi: 10.1136/oemed-2020-107351. Epub 2021 Jul 2. PMID 34215684